CLINICAL TRIAL: NCT00303719
Title: Allogeneic Bone Marrow Transplantation Using Less Intensive Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB Study Closure
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001LS058; UMN-MT2001-10 (Other: Blood and Marrow Transplantation Program); 0108M06725 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma; Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: leukemia; lymphoma; myeloma
MeSH Terms: conditions — Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; fludarabine; fludarabine phosphate; Mycophenolic Acid; Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation; Whole-Body Irradiation; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Risk Patients (Experimental): Nonmyeloablative conditioning using fludarabine, cyclophosphamide and low dose Total Body Irradiation with or without anti-thymocyte globulin followed by allogeneic hematopoietic stem cell transplantation, immunosuppressive cyclosporine and mycophenolate mofetil and post-transplant use of bone marrow-stimulating filgrastim.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine; Drug: mycophenolate mofetil; Procedure: stem cell transplantation; Radiation: total body irradiation; Drug: filgrastim
- Standard Risk Patients (Experimental): Nonmyeloablative conditioning using fludarabine, cyclophosphamide and low dose Total Body Irradiation with or without anti-thymocyte globulin followed by allogeneic hematopoietic stem cell transplantation, immunosuppressive cyclosporine and mycophenolate mofetil and post-transplant use of bone marrow-stimulating filgrastim.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine; Drug: mycophenolate mofetil; Procedure: stem cell transplantation; Radiation: total body irradiation; Drug: filgrastim

INTERVENTIONS:
Biological: anti-thymocyte globulin — ATG dose is 15 mg/kg intravenous (IV) every 12 hours for 6 doses on days -6, -5, and -4.
  Those that should/will receive ATG in the preparative regimen:
  * Related donor recipients who have not had exposure to combination chemotherapy in the 6 months preceding transplant should
  * Unrelated donor recipients who have not had exposure to combination chemotherapy in the 3 months preceding transplant will
  * Unrelated donor recipients who have had only a single induction cycle for the treatment of ALL/AML or MDS or CML blast crisis should
  * Recipients with a prior autologous transplant in the year prior to second transplant do not require ATG.
  Other Names: ATG
Drug: cyclophosphamide — Cyclophosphamide will be given in a two hour infusion, total dose 50 mg/kg on day -6.
  Other Names: Cytoxan
Drug: cyclosporine — Patients will receive cyclosporine A (CSA) therapy beginning on day -3 maintaining a level of >200. For adults the initial dose will be 2.5 mg/kg IV over 2 hours every 12 hours. For children < 40 kg the initial dose will be 2.5 mg/kg IV over 2 hours every 8 hours. Patients will receive CSA until day +100.
  Other Names: CSA
Drug: fludarabine — Fludarabine 30 mg/m^2/day intravenous (IV) on day -6 through day -2., total dose 150 mg/m^2 for 5 days.
  Other Names: Fludara
Drug: mycophenolate mofetil — Mycophenolate mofetil (MMF) 1.5 gram twice a day (BID) or if < 50 kg will be given 15 mg/kg orally(po) BID,beginning on day -3, and discontinue at day +30 or 7 days after engraftment (3 consecutive days of absolute neutrophil count (ANC) > 0.5 x 109 /L).
  Other Names: MMF
Procedure: stem cell transplantation — On day 0, if related donor, stem cells are infused via central line. If unrelated donor, marrow/PBSC is infused after arrival and processing on day 0.
  Other Names: peripheral blood stem cell transplantation; bone marrow transplant
Radiation: total body irradiation — The dose of TBI will be 200 cGy given in a single fraction on day -1.
  Other Names: TBI
Drug: filgrastim — Patients with white blood cell (WBC) counts < 2500 any time after stem cell infusion will be started on G-CSF support at Day +5 at a dose of 5 mcg/kg intravenously or subcutaneously (IV/SQ) daily rounded to vial size until absolute neutrophil count (ANC) > 2500 for 2 consecutive days.
  Other Names: G-CSF

SUMMARY:
RATIONALE: A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and radiation therapy, or that have become cancer. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclophosphamide and fludarabine together with total-body irradiation followed by cyclosporine and mycophenolate mofetil before the transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy together with radiation therapy followed by cyclosporine and mycophenolate mofetil works in treating patients who are undergoing a donor stem cell transplant for hematologic cancer, metastatic breast cancer, or kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if a nonmyeloablative regimen comprising cyclophosphamide, fludarabine, and radiotherapy followed by cyclosporine and mycophenolate mofetil provides a prompt and durable donor engraftment in patients with hematologic malignancies or kidney cancer who are undergoing allogeneic stem cell transplantation.
* Determine the safety of this nonmyeloablative transplantation regimen in these patients.
* Determine the risk of graft-versus-host-disease in patients treated with this regimen.
* Determine the antineoplastic potency of nonmyeloablative stem cell transplantation in patients treated with this regimen.
* Determine the effect of lower doses of daily fludarabine on treatment-related mortality (TRM) OUTLINE: Patients are stratified according to risk (standard vs high).
* Preparative regimen*: Patients receive cyclophosphamide intravenously (IV) over 2 hours on day -6 and fludarabine IV over 1 hour on days -6 to -2. Patients undergo total body irradiation on day -1. Some patients also receive anti-thymocyte globulin (ATG)** IV every 12 hours on days -6 to -4. Patients who receive ATG* include the following:

  * Related donor recipients who have not received combination chemotherapy within the past 6 months
  * Unrelated donor recipients who have not received combination chemotherapy within the past 3 months
  * Unrelated donor recipients who have received only 1 induction course for the treatment of acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), myelodysplastic syndromes (MDS), or blastic phase chronic myelogenous leukemia (CML) NOTE: **Patients who underwent prior autologous stem cell transplantation in the past year do not receive ATG.
* Allogeneic peripheral blood stem cell transplantation (PBSCT): Patients undergo allogeneic PBSCT on day 0.
* Graft-versus-host-disease prophylaxis: Patients receive cyclosporine IV over 2 hours beginning on day -3 and continuing until at least day 100. Patients also receive mycophenolate mofetil IV or orally twice daily on days -3 to 30.
* Donor lymphocyte infusion (DLI): Patients without active GVHD but deteriorating donor chimerism may receive DLI IV over 2 hours.

After completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 300 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

Standard patients will be enrolled into Arms 1-6. High risk patients (transplant with aplasia) will be considered separately in Arm 7.

* Age and Graft criteria (all patients)

  * Patient's < or = 75 years old with a 5/6 or 6/6 related donor match are eligible.
  * Patient's < or = 75 years who have a 7-8/8 HLA-A,B,C,DRB1 allele matched unrelated volunteer marrow and/or peripheral blood stem cell (PBSC) donor match are eligible.
* Disease Criteria (standard risk patients)

  * Acute myelogenous leukemia
  * Acute lymphocytic leukemia
  * Chronic myelogenous leukemia all types except blast crisis (note treated blast crisis in chronic phase is eligible).
  * Non-Hodgkins lymphoma (NHL), Hodgkins, chronic lymphocytic leukemia, multiple myeloma demonstrating chemosensitive disease
  * Acquired bone marrow failure syndromes
  * Myelodysplastic syndrome of all subtypes including refractory anemia (RA) or all IPSS categories if severe pancytopenia, transfusion requirements not responsive to therapy, or high risk cytogenetics. Blasts must be less than 5%. If >5% requires therapy (induction or Hypomethylating agents) pre-transplant to decrease disease burden.
  * Renal cell cancer,
  * Chronic myeloproliferative disorder, i.e. myelofibrosis
* Disease Criteria (High risk patients on Arm 7)

  * Patients with refractory leukemia or MDS may be taken to transplant in aplasia after induction or re-induction chemotherapy or radiolabeled antibody. These high risk patients will be analyzed separately in Arm 7.
* Adequate organ function and performance status (all patients)

Exclusion Criteria:

* Pregnancy or breast feeding
* Evidence of HIV infection or known HIV positive serology
* Active serious infection
* Congenital bone marrow failure syndrome
* Previous irradiation that precludes the safe administration of an additional dose of 200 cGy of total body irradiation (TBI)
* Chronic myelogenous leukemia (CML) in refractory blast crisis
* Intermediate or high grade NHL, mantle cell NHL, and Hodgkins disease that is progressive on salvage therapy. Stable disease is acceptable to move forward provided it is non-bulky.
* Multiple Myeloma progressive on salvage chemotherapy.

DONOR ELIGIBILITY

* Related will undergo apheresis - if donor is unable to undergo apheresis, a bone marrow harvest is acceptable; unrelated volunteer donors must be able to undergo bone marrow harvest or apheresis.
* All donors must be able to give informed consent.
* Donors weighing less than 40 kg (children) will need evaluation by a pediatrician for suitability of the apheresis procedure. Informed consent must be obtained from parent or guardian as applicable for minors.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2002-03-26 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Warlick, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Warlick E, Ahn KW, Pedersen TL, Artz A, de Lima M, Pulsipher M, Akpek G, Aljurf M, Cahn JY, Cairo M, Chen YB, Cooper B, Deol A, Giralt S, Gupta V, Khoury HJ, Kohrt H, Lazarus HM, Lewis I, Olsson R, Pidala J, Savani BN, Seftel M, Socie G, Tallman M, Ustun C, Vij R, Vindelov L, Weisdorf D. Reduced intensity conditioning is superior to nonmyeloablative conditioning for older chronic myelogenous leukemia patients undergoing hematopoietic cell transplant during the tyrosine kinase inhibitor era. Blood. 2012 Apr 26;119(17):4083-90. doi: 10.1182/blood-2012-02-409763. Epub 2012 Mar 9. PMID 22408257
- [Background] Warlick ED, DeFor TE, Bejanyan N, Holtan S, MacMillan M, Blazar BR, Dusenbery K, Arora M, Bachanova V, Cooley S, Lazaryan A, McGlave P, Miller JS, Rashidi A, Slungaard A, Vercellotti G, Ustun C, Brunsein C, Weisdorf D. Reduced-Intensity Conditioning Followed by Related and Unrelated Allografts for Hematologic Malignancies: Expanded Analysis and Long-Term Follow-Up. Biol Blood Marrow Transplant. 2019 Jan;25(1):56-62. doi: 10.1016/j.bbmt.2018.07.038. Epub 2018 Aug 1. PMID 30077015
- [Derived] Bachanova V, Burke MJ, Yohe S, Cao Q, Sandhu K, Singleton TP, Brunstein CG, Wagner JE, Verneris MR, Weisdorf DJ. Unrelated cord blood transplantation in adult and pediatric acute lymphoblastic leukemia: effect of minimal residual disease on relapse and survival. Biol Blood Marrow Transplant. 2012 Jun;18(6):963-8. doi: 10.1016/j.bbmt.2012.02.012. Epub 2012 Mar 16. PMID 22430088
- [Derived] Bachanova V, Sandhu K, Yohe S, Cao Q, Burke MJ, Verneris MR, Weisdorf D. Allogeneic hematopoietic stem cell transplantation overcomes the adverse prognostic impact of CD20 expression in acute lymphoblastic leukemia. Blood. 2011 May 12;117(19):5261-3. doi: 10.1182/blood-2011-01-329573. Epub 2011 Mar 14. PMID 21403127
- [Derived] Bachanova V, Verneris MR, DeFor T, Brunstein CG, Weisdorf DJ. Prolonged survival in adults with acute lymphoblastic leukemia after reduced-intensity conditioning with cord blood or sibling donor transplantation. Blood. 2009 Mar 26;113(13):2902-5. doi: 10.1182/blood-2008-10-184093. Epub 2009 Jan 28. PMID 19179301
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6310652/

RESULTS

PARTICIPANT FLOW:
Groups:
- High Risk Patients: Patients with refractory leukemia or MDS
- Standard Risk Patients: Patients with Disease criteria: Acute myelogenous leukemia , Acute lymphocytic leukemia, Chronic myelogenous leukemia , NHL, Hodgkins, chronic lymphocytic leukemia, multiple myeloma, Acquired bone marrow failure syndromes, Myelodysplastic syndrome, Renal cell cancer,Chronic myeloproliferative disorder
Period: Overall Study
Arm/Group | High Risk Patients | Standard Risk Patients
Started | 13 | 329
Completed | 13 | 292
Not Completed | 0 | 37
Not completed — Not evaluable, prior therapies | 0 | 30
Not completed — Lost to Follow-up | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk Patients | Standard Risk Patients | Total
Number analyzed (Participants) | 13 | 292 | 305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 184 | 188
  >=65 years | 9 | 108 | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 112 | 116
  Male | 9 | 180 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 10 | 250 | 260
  Unknown or Not Reported | 2 | 39 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 12 | 259 | 271
  More than one race | 0 | 6 | 6
  Unknown or Not Reported | 1 | 16 | 17

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil and Donor Cell Engraftment
Description: Successful sustained engraftment is defined as primary neutrophil engraftment by day 42 and e90% donor cells at day 100, with or without DLI.
  Engraftment based on absolute neutrophil count of donor origin > 0.5 x 10e9 /L for 3 days by day 42
Time Frame: Day 42 and Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Patients | Standard Risk Patients
Number analyzed (Participants) | 13 | 292
Participants | 12 | 289

2. Secondary Outcome: Serious Adverse Events
Description: Safety by development of severe adverse events within 100 days of transplant
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Patients | Standard Risk Patients
Number analyzed (Participants) | 13 | 292
Participants | 0 | 47

3. Secondary Outcome: Transplant Related Mortality
Description: > 30% transplant related mortality at 100 days (non-relapse).
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Groups:
- Standard Risk Patients: Patients with Disease criteria: Acute myelogenous leukemia , Acute lymphocytic leukemia, Chronic myelogenous leukemia , NHL, Hodgkins, chronic lymphocytic leukemia, multiple myeloma, Acquired bone marrow failure syndromes, Myelodysplastic syndrome,Chronic myeloproliferative disorder
Arm/Group | High Risk Patients | Standard Risk Patients
Number analyzed (Participants) | 13 | 292
Participants | 2 | 40

4. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Patients | Standard Risk Patients
Number analyzed (Participants) | 13 | 292
Participants | 8 | 181

5. Secondary Outcome: Acute Graft-Versus-Host Disease
Description: Grade III-IV graft versus host disease
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Patients | Standard Risk Patients
Number analyzed (Participants) | 13 | 292
Participants | 2 | 79

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | High Risk Patients | Standard Risk Patients
All-Cause Mortality (participants affected / at risk) | 6/13 | 124/292
Serious Adverse Events (participants affected / at risk) | 1/13 | 53/292
Other Adverse Events (participants affected / at risk) | 12/13 | 272/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Patients (N=13) | Standard Risk Patients (N=292)
Graft versus Host disease (Immune system disorders) | 0 | 28
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 21
Infection (Infections and infestations) | 0 | 4
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk Patients (N=13) | Standard Risk Patients (N=292)
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 17 (18)
Bacterial infection (Infections and infestations) | 5 (15) | 128 (334)
Bleeding (Gastrointestinal disorders) | 2 (4) | 45 (56)
Cystitis (Renal and urinary disorders) | 1 (1) | 15 (18)
Hemodialysis (Renal and urinary disorders) | 2 (2) | 18 (21)
Infection (Etiology unknown) (Infections and infestations) | 4 (8) | 96 (219)
Organ failure (Cardiac disorders) | 2 (4) | 17 (21)
Fungal infection (Infections and infestations) | 4 (15) | 122 (269)
Neuropathy (Nervous system disorders) | 1 (1) | 43 (51)
Neurotoxicity (Nervous system disorders) | 0 (0) | 29 (37)
perihilar opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (20)
Other disorders (General disorders) | 9 (25) | 179 (489)
Pnemonia (Infections and infestations) | 8 (15) | 149 (351)
Ear disorder (Ear and labyrinth disorders) | 2 (2) | 10 (10)
Increased oxygen requirement (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 61 (73)
Viral infection (Infections and infestations) | 8 (15) | 143 (291)
Abnormal liver (Hepatobiliary disorders) | 0 (0) | 18 (20)
Decrease cardiac function (Cardiac disorders) | 0 (0) | 28 (33)
pericardial effusion (Cardiac disorders) | 2 (3) | 45 (51)
Eye disorder (Eye disorders) | 0 (0) | 31 (48)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT00303719/Prot_SAP_000.pdf